CLINICAL TRIAL: NCT03504189
Title: Clinical Study Evaluating the Safety of PregSense and Comparative Performance of PregSense Versus CTG in Prenatal Monitoring of Pregnant Subjects
Brief Title: Evaluating the Safety of PregSense™ and Compare Its Performance to CTG in Prenatal Monitoring of Pregnant Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuvo-Group, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLP1000
Record Dates: First submitted 2018-03-05; First posted 2018-04-20 (Actual); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy
Keywords: Fetal monitoring, Prenatal monitoring

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PregSense™ (Experimental): PregSense™ wearable device and the standard of care CTG (cardiotocography) will be applied for maternal-fetal monitoring
  Interventions: Device: PregSense™; Device: Cardiotocopraphy (CTG)

INTERVENTIONS:
Device: PregSense™ — PregSense™ wearable device will be applied for maternal-fetal monitoring
Device: Cardiotocopraphy (CTG) — Cardiotocopraphy (CTG) will be applied for maternal-fetal monitoring

SUMMARY:
This clinical study will evaluate the safety of PregSense™ and Comparative Performance of PregSense™ versus CTG in Prenatal Monitoring of Pregnant subjects.

DETAILED DESCRIPTION:
PregSense™ is a maternal-fetal monitor that non-invasively measures and displays fetal heart rate, maternal hear rate and uterine contractions. This study will be performed to collect and digitally record data from PregSense™ and the standard of care (CTG) in order to provide evidence of safety and agreement between PregSense™ and the gold standard NST device.

ELIGIBILITY:
Inclusion Criteria:

* Female age between 18-50
* Gestational age > 32 + 0 weeks
* Singleton gestation
* Ability to understand and sign informed consent

Exclusion Criteria:

* BMI (Body Mass Index) ≥ 45 and ≤15 prior pregnancy
* Multiple gestation
* Uncontrolled Hypertension
* Fetal Anomaly
* Subjects with skin problems in the abdominal area (such as flesh wounds, cuts in the skin, skin rashes, etc.)
* Subjects with implanted electronic devices (pacemaker, defibrillator, etc.)
* Subjects who, in the judgement of the investigator, are likely to be non-compliant or uncooperative during the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 151 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia
- Heidelberg University Womens Hospital, Heidelberg, Germany
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mhajna M, Schwartz N, Levit-Rosen L, Warsof S, Lipschuetz M, Jakobs M, Rychik J, Sohn C, Yagel S. Wireless, remote solution for home fetal and maternal heart rate monitoring. Am J Obstet Gynecol MFM. 2020 May;2(2):100101. doi: 10.1016/j.ajogmf.2020.100101. Epub 2020 Mar 17. PMID 33345967

RESULTS

PARTICIPANT FLOW:
Groups:
- "PregSense™ and Cardiotocopraphy (CTG)": PregSense™ WSB then was applied by the authorized study personnel to the maternal abdominal area, not before cleaning the maternal abdomen with a damp cloth, then drying the abdomen. Before initiating the recording session, a valid signal is to be obtained.
  An authorized study personnel applied the CTG transducers and confirmed fetal heart rate detection according to the standard of care procedure.
  If a valid signal was detected, a 30-minute session initiated, recording both systems simultaneously in a synchronized method (PregSense™ and CTG).
  Following the completion of the sessions, the authorized study personnel removed both monitoring systems from the maternal abdomen.
Period: Overall Study
Arm/Group | "PregSense™ and Cardiotocopraphy (CTG)"
Started | 151
Completed | 147
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Screening Failure | 1
Not completed — Device Failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | PregSense™
Number analyzed (Participants) | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 147
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 140
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69
  Israel | 49
  Germany | 31

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate
Description: Provide evidence of safety and FHR agreement between PregSense™ and the standard of care devices (i.e. CTG)
Time Frame: 30 Minutes
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- "PregSense™ and Cardiotocopraphy (CTG)": PregSense™ wearable device was applied for maternal-fetal monitoring
- Cardiotocopraphy (CTG): Philips FM30 (CTG) was applied for maternal-fetal monitoring
Arm/Group | "PregSense™ and Cardiotocopraphy (CTG)" | Cardiotocopraphy (CTG)
Number analyzed (Participants) | 147 | 147
bpm | 140.3 (11.9) | 140.4 (11.65)

2. Primary Outcome: Maternal Heart Rate
Description: Provide evidence of safety and agreement between MHR collected via the PregSense™ and the standard of care devices (i.e. CTG)
Time Frame: 30 MInutes
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- PregSense™: PregSense™ wearable device was applied for maternal-fetal monitoring
- Cardiotocopraphy (CTG): Philips FM30 Cardiotocopraphy (CTG) was applied for maternal-fetal monitoring
Arm/Group | PregSense™ | Cardiotocopraphy (CTG)
Number analyzed (Participants) | 147 | 147
bpm | 89.3 (12.54) | 89.1 (12.5)

3. Secondary Outcome: Uterine Contractions
Description: Compare uterine contractions from Pregsense™ versus CTG.
Time Frame: 30 Minutes
Population: Uterine Contraction information was eventually not collected AT ALL, therefore no population to describe.
Groups:
- "PregSense™ and Cardiotocopraphy (CTG)": PregSense™ wearable device and the standard of care CTG (cardiotocography) will be applied for maternal-fetal monitoring
  PregSense™: PregSense™ wearable device will be applied for maternal-fetal monitoring
  Cardiotocopraphy (CTG): Cardiotocopraphy (CTG) will be applied for maternal-fetal monitoring
Arm/Group | "PregSense™ and Cardiotocopraphy (CTG)"
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Safety Measures
Description: Evaluate device related adverse events
Time Frame: Through study completion, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | PregSense™
Number analyzed (Participants) | 147
Participants | 0

ADVERSE EVENTS:
Time Frame: 30 minutes during Non stress test (NST)
Description: No adverse events reported during the trial
Arm/Group | PregSense™
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 0/147

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03504189/Prot_SAP_000.pdf